CLINICAL TRIAL: NCT05954936
Title: Trauma Registry in a General Hospital From Villavicencio, Colombia, First Semester 2023: An Observational Retrospective Trial
Brief Title: Trauma Registry in Villavicencio, Colombia
Acronym: TRaVi
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Principal investigator, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2023_02_TRAUMA
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Trauma; Trauma Blunt; Penetrating Wounds; Severe Trauma; Polytrauma; Registries
Keywords: Wounds and Injuries; Trauma Severity Indices; Trauma Centers; Multiple Trauma; Registries; Data Collection; Routinely Collected Health Data; Colombia
MeSH Terms: conditions — Wounds and Injuries; Wounds, Nonpenetrating; Wounds, Penetrating; Multiple Trauma | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blunt injury: Patients with non-penetrating injuries from falls, car accidents, or other mechanisms. Injuries that were caused by impact with a blunt object where there is no penetration of the skin.
  Interventions: Other: Risk factor
- Penetrating injury: Penetrating wounds by guns, knives, and other penetrating injuries. Wounds that were caused by objects penetrating the skin.
  Interventions: Other: Risk factor

INTERVENTIONS:
Other: Risk factor — No therapeutic or diagnostic intervention will be provided; it is an observational study.

SUMMARY:
Introduction: Injuries are a leading cause of mortality worldwide. It is necessary to know the incidence of injuries, mechanisms of wounds, therapy provided, and outcomes. Trauma registries are useful to describe the population served in specialized centers. Nevertheless, it is necessary also to identify the peculiarities of the event in the province and institutions non-dedicated to trauma attention.

Objective: The study aims to describe the initial experience with a trauma register in a general hospital in the Colombian Orinoquia.

Methodology: The investigators designed an observational retrospective study to analyze the admission database and revision of history charts of patients older than 15 years admitted for trauma from January to June 2023 in a hospital from Villavicencio, Colombia. The information will be exported to Excel for debugging and analysis. A description of the frequency and proportion of categorical variables will be performed; the central distribution and dispersion of quantitative variables will be reported. U of Mann-Whitney and Chi-square tests will be used to compare the variables by outcome; a p<0.05 was selected as a significant value.

Conclusions: It will be a pioneer study in this region, and it is necessary to evaluate the incidence of patients admitted by trauma, the mechanisms and type of injury, the care provided, and the outcomes.

DETAILED DESCRIPTION:
Trauma is a leading cause of global mortality or incapacitation in survivors. The population involved is mainly young adult men affected by preventable injuries. Knowing the incidence of injuries, mechanisms of wounds, approaching strategies, and outcomes is essential to review individual interventions and collective policies to improve prevention.

Casualties in Colombia had a high incidence in previous decades; injuries and attributable deaths have recently decreased, but they are still the third cause of mortality. Contrary to high-income countries, interpersonal violence is the predominant mechanism involved.

Data registries are used worldwide in specialized centers that focus on providing healthcare in trauma. Nevertheless, it is necessary also to know the incidence in community and non-dedicated general hospitals.

Determining the characteristics of patients admitted to the emergency ward by injuries will provide essential information on the severity, mechanisms, type of population affected, immediate or consequential care delivered, and outcomes. Such an analysis will give knowledge to prioritize policies, resources, upgrade clinical practice guidelines, and improve results.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency ward by trauma.

Exclusion Criteria:

* None.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The trial participants are those admitted requesting emergency attention by trauma during the study period, according to the registers of admission in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients dead | 28 days or discharge
  Mortality on discharge or the first 28 days of hospitalization

SECONDARY OUTCOMES:
Number of days in hospitalization | 28 days or discharge
  Hospital length of stay
Number of patients needing ICU | 28 days or discharge
  Need of ICU
Number of days in ICU | 28 days or discharge
  ICU length of stay
Number of patients needing mechanical ventilation | 28 days or discharge
  Need of mechanical ventilation
Number of days in mechanical ventilation | 28 days or discharge
  Length of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Cooperative University of Colombia
Locations (1):
- Clinica Primavera, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
Database will not be shared to provide confidentiality to the identity of patients.

REFERENCES:
- [Result] Ordonez CA, Morales M, Rojas-Mirquez JC, Bonilla-Escobar FJ, Badiel M, Minan Arana F, Gonzalez A, Pino LF, Uribe-Gomez A, Herrera MA, Gutierrez-Martinez MI, Puyana JC, Abutanos M, Ivatury RR. Trauma Registry of the Pan-American Trauma Society: One year of experience in two hospitals in southwest Colombia. Colomb Med (Cali). 2016 Sep 30;47(3):148-154. PMID 27821894
- [Result] Uribe A, Ordóñez CA, Badiel M, Tejada JW, Harry Loaiza J, Fernando Pino L, et al. Tendencia del trauma en dos hospitales nivel IV en Cali, Colombia. Reporte preliminar en la Plataforma del Registro de la Sociedad Panamericana de Trauma (SPT/RT). Panam J Trauma Crit Care Emerg Surg. 2012;1(3):175-81.
- [Result] Christey G, Warren J, Palmer CS, Burrell M, Vallmuur K. Development of a standardized minimum dataset for including low-severity trauma patients in trauma registry collections in Australia and Aotearoa New Zealand. ANZ J Surg. 2023 Mar;93(3):572-576. doi: 10.1111/ans.18326. Epub 2023 Mar 1. PMID 36856198
- [Result] Ordóñez CA, Botache WF, Pino LF, Badiel M, Tejada JW, Sanjuán J, et al. Experiencia en dos hospitales de tercer nivel de atención del suroccidente de Colombia en la aplicación del Registro Internacional de Trauma de la Sociedad Panamericana de Trauma. Rev Colomb Cir. 2013;28(1):39-47.
- [Result] Eyler L, Hubbard A, Juillard C. Assessment of economic status in trauma registries: A new algorithm for generating population-specific clustering-based models of economic status for time-constrained low-resource settings. Int J Med Inform. 2016 Oct;94:49-58. doi: 10.1016/j.ijmedinf.2016.05.004. Epub 2016 Jun 29. PMID 27573311
- [Result] Carius BM, Bebarta GE, April MD, Fisher AD, Rizzo J, Ketter P, Wenke JC, Salinas J, Bebarta VS, Schauer SG. A Retrospective Analysis of Combat Injury Patterns and Prehospital Interventions Associated with the Development of Sepsis. Prehosp Emerg Care. 2023;27(1):18-23. doi: 10.1080/10903127.2021.2001612. Epub 2021 Dec 22. PMID 34731068
- [Result] Arbizu-Fernandez E, Echarri-Sucunza A, Galbete A, Fortun-Moral M, Belzunegui-Otano T. Epidemiology of severe trauma in Navarra for 10 years: out-of-hospital/ in-hospital deaths and survivors. BMC Emerg Med. 2023 May 24;23(1):54. doi: 10.1186/s12873-023-00818-6. PMID 37226131
- [Result] Mandavia D, Newton K. Geriatric trauma. Emerg Med Clin North Am. 1998 Feb;16(1):257-74. doi: 10.1016/s0733-8627(05)70358-8. PMID 9496324
- [Result] Cleves D, Gomez C, Davalos DM, Garcia X, Astudillo RE. Pediatric trauma at a general hospital in Cali, Colombia. J Pediatr Surg. 2016 Aug;51(8):1341-5. doi: 10.1016/j.jpedsurg.2016.01.008. Epub 2016 Feb 3. PMID 26879744
- [Result] Benjamin ER, Demetriades D, Owattanapanich N, Shackelford SA, Roedel E, Polk TM, Biswas S, Rasmussen T. Therapeutic Interventions and Outcomes in Civilian and Military Isolated Gunshot Wounds to the Head: A Department of Defense Trauma Registry and ACS TQIP-matched Study. Ann Surg. 2023 Jul 1;278(1):e131-e136. doi: 10.1097/SLA.0000000000005496. Epub 2022 Jul 4. PMID 35786669
- [Result] Fitschen-Oestern S, Lippross S, Lefering R, Kluter T, Weuster M, Franke GM, Kirsten N, Muller M, Schroder O, Seekamp A; TraumaRegister DGU. Does the time of the day affect multiple trauma care in hospitals? A retrospective analysis of data from the TraumaRegister DGU(R). BMC Emerg Med. 2021 Nov 13;21(1):134. doi: 10.1186/s12873-021-00525-0. PMID 34773984